CLINICAL TRIAL: NCT04308213
Title: Interventional Study on the Treatment of Shoulder Osteoarthritis With Intra-articular Injections of Autologous Bone Marrow Aspirate.
Brief Title: Study on Shoulder Arthritis Treatment With Intra-articular Injections of Autologous Bone Marrow Aspirate.
Acronym: Stemshoulder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 955
Record Dates: First submitted 2020-03-10; First posted 2020-03-13 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Shoulder Arthritis
Keywords: arthritis; mesenchymal stem cells
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bone Marrow aspirate (Experimental): All the patients enrolled in the study will be treated with the bone marrow aspirate obtained with the Bone Marrow Cellution Kit.
  Interventions: Device: Marrow Cellution System

INTERVENTIONS:
Device: Marrow Cellution System — The treatment will be carried out in the operating room under ordinary hospitalization and provides the intra-articular application of 9 ml of autologous bone marrow aspirate in the glenohumeral joint affected by arthrosis. To obtain the necessary amount, a bone marrow aspirate of about 12 ml will be taken from the iliac crest by means of the Marrow Cellution System, Geistlich Italia. This autologous bone marrow aspirate will be injected using the same syringe into the glenohumeral joint affected by arthrosis under amplioscopic control.

SUMMARY:
Treatment of isolated osteoarthritis of the glenohumeral joint at the initial stages involves the use of numerous conservative or arthroscopic treatments with uncertain results and, upon their failure, the current solution for the resolution of symptoms is shoulder arthroplasty, an effective procedure but with significant costs and rates of morbidity, especially in young patients. Since the use of intra-articular injections of mesenchymal cells obtained from the bone marrow has proved effective in the treatment of gonarthrosis, our goal is to evaluate the effectiveness of the same therapy in the treatment of glenohumeral arthritis isolated.

DETAILED DESCRIPTION:
Glenohumeral arthritis is one of the main reasons for persistent shoulder pain and reduced movement (range of motion, ROM) as it can compromise the work activity and also the normal daily activities, leading to the development of depressive syndromes. The final treatment is shoulder arthroplasty, which is effective but is associated with significant costs and morbidity rates. In addition, arthro-prosthesis is avoided in young patients due to longevity concerns and is not indicated in the early stages of arthritis. Currently, conservative treatments for patients with mild or moderate glenohumeral arthritis include non-steroidal anti-inflammatory drugs (NSAIDs), corticosteroid injections, with low efficacy and a significant adverse effect profile, hyaluronic acid infiltrations, with good efficacy in initial treatment, and infiltrations of platelet-Rich Plasma (PRP), which have shown beneficial effects in knee arthritis. However, evidence for the glenohumeral joint are limited. In cases not responsive to conservative therapy, and especially in young patients, a valid alternative to the prosthesis is the arthroscopic treatment, with good results in the short term, but with relatively high failure rates that increase over time. Other types of nonprosthetic surgical treatment for chondral-humeral defects have low scientific evidence, with variable and uncertain results. In recent years, mesenchymal stem cells (MSC), derived from bone marrow or adipose tissue, due to the ability to differentiate into chondrogenic line cells, have emerged as cells with great therapeutic potential in patients with degenerative joint disorders. Since the knee joint is the most susceptible to pathology because of its mechanical load, most studies based on stem cell therapy regard the knee joint, reporting promising results in treatment in the treatment of early stages of arthritis. As regards the glenohumeral joint, since the most frequent pathology affects the tendons of the rotator cuff, almost all studies investigate the effect of MSC in the treatment of rotator cuff disorders with or without associated surgical repair techniques. Only a prospective study analyzed the effect of intra-articular MSC injection derived from bone marrow in 34 patients with isolated glenohumeral arthritis, reporting a significant decrease in pain and an improvement in shoulder function measured by the Disabilities of the Arm, Shoulder and Hand (DASH) scale at about 1 year, although study quality is very low. Since the use of intra-articular injections of mesenchymal cells obtained from the bone marrow has proved effective in the treatment of gonarthrosis, our study proposes to evaluate the long-term efficacy of this type of therapy in the treatment of the isolated glenohumeral arthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged between 35 and 75.
2. Light or moderate glenohumeral arthritis assessed by MRI.
3. Failure after at least 6 months of conservative treatment (patients not responding to drug therapy with NSAIDs and pain killers, no benefit from hydro-kinesitherapy or physiotherapy, no benefit after a course of hyaluronic acid or PRP infiltrations, or after at least one corticosteroid infiltration)
4. Ability and consent of patients to participate actively in the rehabilitation and clinical and radiological follow-up protocol;
5. The signing of informed consent.

Exclusion Criteria:

1. Patients incapable of understanding and will
2. Patients with shoulder trauma within 6 months prior to surgery
3. Patients with malignancies;
4. Patients with rheumatic diseases;
5. Patients with diabetes;
6. Patients with metabolic thyroid disorders;
7. Patients abusing alcoholic beverages, drugs or drugs;
8. Patients with signs of rotator cuff or long head biceps disease at MRI
9. Patients with a history of untreated shoulder instability.
10. Patients with arthroscopic evidence of rotator cuff injuries.
11. Glenohumeral arthrosis "bone to bone".

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-11-12 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Change of the Constant-Murley score | Timepoints: Screening, 3, 6, 12, 24, 36, and 48 months
  Constant-Murley score: is a scale of 100 points that defines the level of pain and the ability to perform normal daily activities of the patient. The test is divided into 4 subscales: pain (15 points), daily life activity (20 points), force (25 points), range of movement: forward elevation, external rotation, abduction and internal rotation of the shoulder (40 points).
Change of the VAS pain score | Timepoints: Screening, 3, 6, 12, 24, 36, and 48 months
  Visual analogue Scale (VAS): The patient is asked to quantify pain by indicating its intensity on an visual analog scale (0 no pain, 10 the worst pain).

SECONDARY OUTCOMES:
Change of range of motion (ROM) | Timepoints: screening, 6, 12, 24, 36 and 48 months
  Range of motion (ROM): the range of motion will be evaluated during the clinical examination using a goniometer in terms of anterior flexion, abduction, external rotation with elbow to side (ER1), external rotation with elbow abducted to 90° (ER2) and internal rotation (level reached with the hand on the back).
clinical change based on the DASH scale (disability of the arm, shoulder and Hand) | Timepoints: screening, 6, 12, 24, 36 and 48 months
  DASH (Disabilities of the arm, shoulder and Hand) rating card: is a questionnaire that asks to evaluate the difficulty in carrying out 30 daily tasks, bringing a score from 0 (best functionality) to 100 (worst functionality).
clinical change based on the , American Shoulder and Elbow Surgeons (ASES) score | Timepoints: screening, 6, 12, 24, 36 and 48 months
  ASES (American shoulder and Elbow Surgeons shoulder Score) rating card: questionnaire that integrates the pain felt (rated on a scale of 0 to 10) and the ability to perform 10 daily activities in which the use of the arm is involved, reporting a score from 0 (worst functionality) to 100 (best functionality).
evaluation of shoulder MRI results | 12 and 24 months
  Execution of a shoulder MRI for evaluation of joint cartilage by comparing it with the MRIs of previous time points.
evaluation of shoulder X-ray (XR) results | 12, 24 and 48 months
  Execution of a shoulder XR in antero-posterior (AP) projection to assess the progression of glenohumeral arthrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Castagna, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No